CLINICAL TRIAL: NCT05879900
Title: Effects of a Fifteen-minute Functional Exercise Intervention on Levels of Physical Fitness of Schoolchildren
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Gabriel Gustavo Bergmann, Principal Investigator, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESEF-UFPel
Record Dates: First submitted 2023-05-06; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Physical Fitness
Keywords: Physical Fitness; Physical Activity; Schools; Physical Education and Training; Intervention Study
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The research methodology consists of 230 participants, of which 115 subjects will be the Control Group with interventions to be carried out: pre and post-intervention measures and the other 115 subjects will be the Intervention Group with interventions of pre- and post-intervention measures, and participation of the study intervention.
Who Masked: Outcomes Assessor
Masking Description: The blinding process will only be in relation to the evaluators of the pre- and post-intervention variables and those responsible for the tabulation and data analysis. Regarding the blinding of the sample and teachers participating in the intervention, it will not be possible to blind the process of clarity and understanding of the intervention in which the group will participate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - IG (Experimental): The intervention group will have in their Physical Education classes the inclusion of functional physical exercises lasting approximately 15 minutes at the beginning of the classes. After the intervention, the classes will continue according their previously planned contents. Classes take place twice a week, on non-consecutive days. In this way, the intervention program will take place over 12 weeks, totaling 24 sessions distributed in 24 classes. The exercises will be performed with natural body movements such as running, jumping, jumping, pulling, crouching, turning and pushing in order to develop Physical Fitness. During the intervention program period there will be an increase in intensities and complexity going through processes that follow the initial, intermediate and final preparation and progression.
  Interventions: Other: Functional physical exercises
- Comparator Group - CG (Active Comparator): The comparator group wil keep performing the Physical Education classes according their previously planned contents.
  Interventions: Other: Physical Education classes

INTERVENTIONS:
Other: Functional physical exercises — Functional physical exercises lasting approximately 15 minutes, for 12 weeks or 24 sessions. The exercises take place during physical education classes taught by the physical education teachers in charge of the classes. The place of intervention takes place in full-time schools in the rural area.
  Arms: Intervention Group - IG
Other: Physical Education classes — Physical Education classes according their previously planned contents.
  Arms: Comparator Group - CG

SUMMARY:
This is an intervention research project, with a pragmatic experimental design of the type Randomized Clinical Trial. Schoolchildren from 6th to 9th grade of both genders, adolescents must be in age group between 10 and 17 years old. enrolled in public schools in the city of Canguçu/RS in the rural zone full-time that have professors with academic training in the area of EF will be allocated in intervention group (IG) and control group (CG). The GI will participate in the inclusion of 15 minutes of functional exercises during the PE class and the GC will continue with the PE classes as planning elaborated by the teachers and pedagogical coordination. The study variables will be organized into main dependents (physical parameters related to health), secondary dependents (parameters behavioral and psychological health-related), characterization of the participants, and independent.

After the 12 weeks of intervention, the data will be collected again, in order to compare the data obtained before the intervention. The expected results after 12 weeks will be that the Group intervention has a significant improvement in the physical, behavioral and psychosocial parameters of health compared to the control group.

DETAILED DESCRIPTION:
1. OBJECTIVES

   General:

   As a general objective to evaluate the effects of a fifteen-minute intervention of functional exercises during PE classes on physical, behavioral and psychosocial health parameters in schoolchildren.

   Specific:

   Check the effects of the intervention with fifteen-minute functional exercises:
   * In cardiorespiratory fitness
   * In strength, endurance and muscle power
   * On speed and agility
   * On flexibility
   * On body mass index, waist circumference and skinfolds
   * In physical activity levels
   * In recreational screen time
   * In self-concept
   * Motivation for participation in PE classes
   * In mental health (symptoms of stress, anxiety and depression).
2. STUDY METHODOLOGY

   The Study consists of 230 participants, with 115 subjects being the Control Group (GC) with interventions to be carried out: pre and post-intervention measures and the other 115 subjects will be the Intervention Group (IG) with interventions of pre- and post-intervention measures, and participation of the study intervention.

   Contact was made with the management teams of the schools to present the study proposal, as well as as the request for its realization in the dependencies of the schools. With the authorization of SMEEC and directive teams, the Physical Education teachers responsible for the schools in the final years of elementary school were contacted and the project objectives presented. It was also explained that the teachers who make up the GI will participate in training to apply the training program intervention and that the teachers who make up the GC will be offered the same training at the end of the study. In each EDUCCAN there is a Physical Education teacher.

   Thus, among the teachers who expressed interest and consented to participate in the study, all professors, internal (titular) or external, signed a Term of Free and Informed Consent (TCLE) signaling your acceptance to participate in the study.

   There was a simple raffle dividing them into groups that received training to apply the training program intervention before the beginning of the study (teachers who composed the IG) and after the end of the study (teachers who may compose the GC).

   The teachers drawn to compose the GC were invited to participate in a training course on Sports Praxeology in the same period of formation of the GI. After intervention, the GI was invited to participate in training on Sports Praxeology and the GC in training on the functional exercise intervention. Allocation of Groups The process of allocation of groups took place in the following way: EDUCCANs Physical Education teachers (graduated in PE) who agreed to participate in the study were drawn to participate in training on the intervention program before the start of the study (the teachers who made up the GI) and after the end of the study (teachers who made up the CG). The teachers who were drawn to the GI participated in training on the intervention program before the start of the study and are responsible for carrying out the intervention activities of this project. The students of classes in the final years of elementary school in the schools where these teachers work were invited to participate in the intervention. GC teachers participated in training on Praxeology Sports and were instructed to keep their classes according to the planning previously carried out by them following the SMEEC guidelines. It is noteworthy that the GC professors will be invited to participate in the same IG training after the end of the intervention period.

   The number of teachers who had their classes evaluated participating in the study was defined according to the number of students enrolled per school where these teachers work. Thus, among teachers who agreed to participate in the study, a simple drawing was carried out. Initially, a teacher was drawn who participated in the training (GI) and the number of students enrolled in the school where this teacher teaches. The number of drawn teachers was defined considering the estimated number of students to compose the IG and GC, according to the sample size calculation. The same procedure was carried out in relation to the teachers who participated in the training only after the completion of the study and, therefore, it will be the teachers of the classes that will form the GC.

   The training of school teachers (EDUCCAN) was conducted by the teachers responsible for project and was carried out in a hybrid and face-to-face manner. The teachers that intervention applicators are physical education teachers trained in the area and full professors of the classes. The pre- and post-intervention measures are carried out by an evaluation team made up of students and professors from the field of physical education. The evaluation team went through face-to-face theoretical-practical training on the procedures and standardization for applying the evaluative instruments aimed at pre and post intervention tests.

   The variables and measurement procedures of the study were organized into main dependents (physical parameters related to health), secondary (behavioral and psychological parameters related to health), characterization of participants, and independent. Main Dependent Variables The physical parameters related to the analyzed will be: Anthropometric Indicators, Cardiorespiratory Fitness (APC), Strength/Endurance Muscle (FRM), Handgrip Strength, Power of Lower Limbs, Speed, Agility and Flexibility (FLEX). Anthropometric Indicators The anthropometric indicators analyzed will be the height (cm), body mass (kg), waist circumference (cm), sitting height (cm), and skinfolds triceps and subscapular skin (mm).

   The evaluations will be carried out using the classroom space, during one of the Education classes Physics of selected schools. The teachers, accompanied by the team of evaluators responsible application, they must complete the instrument (Questionnaire) by themselves, requesting support in case of doubt. Anthropometric measurements and physical fitness tests were also applied in the week before the interventions using a second moment of one of the discipline's classes. To the height and body mass measurements will be carried out in a reserved room made available by the directions of schools. Physical fitness tests will be carried out in the space intended for Education classes Physics from both schools. That same week, in the classroom, a familiarization will be proposed in in relation to the subjective perception of Borg Effort scale for students belonging to the intervention with functional cardiorespiratory and strength exercises. Finally, the collections will be carried out again in both schools in the subsequent week after the end of the interventions, using the same logistics of the initial data collection. Description of the intervention Intervention Group (IG) Students who composing the intervention group will have in their PE classes the inclusion of functional physical exercises about 15 minutes of class. After the intervention, the classes continue with their pre-planned content. At EDUCCAN there are three PE periods/classes per week with 50 minutes long each.

   The structuring comprises a 12-week intervention or 24 classes.
3. STATISTICAL ANALYSIS

   The data will be double typed in the EpiData 3.1 software, exported and analyzed using the statistical package SPSS version 20.0. Initially numerical variables will be analyzed in relation to the normality of their distributions using the Shapiro-Wilk test. The description of numerical variables will be performed by mean (x) and standard deviation (sd) or median and interquartile differences. The description of categorical variables will be carried out by absolute (n) and relative (%) frequencies.

   To compare the characterization variables between the groups, the t test for independent samples and the chi-square test for numerical and categorical variables, respectively, will be used. Generalized Estimating Equations (GEE) and Bonferroni's post-hoc test will be used to compare time points (pre and post-intervention) between groups and to identify the group*time interaction.

   The amplitude of the effect sizes will be verified through Cohen's "d", obtaining the classification: small effect size (0.20 to 0.49); medium (0.50 to 0.79); large (0.80 to 1.29); very large (≥1.30), according to (ROSENTHAL, 1996).

   Analyzes will be performed by intention to treat and by protocol. In intention-to-treat analyses, all participants will be included. In the analyzes per protocol, participants who did not present consistent data in at least one of the moments (pre and/or post-intervention) and those who did not participate in at least 75% of the classes will be removed. The significance level adopted will be 5% for all statistical analyses.
4. ETHICAL ASPECTS

By complying with the ethical requirements of the research, the project was qualified and the necessary adjustments were made as suggested by the opinion of the qualification board, later it was submitted via Plataforma Brasil to the Ethics Committee in Research for Human Beings of the Higher School of Physical Education of the Federal University of Pelotas (ESEF/UFPel) and approved according to protocol 66152922.7.0000.5313 following all ethical principles involving human beings to carry out this study.

The participants, parents and/or legal guardians were duly informed about the objectives and procedures of the study through the Free and Informed Assent Term (TALE) of the minor signed by the students participating in the research and the legal guardians of the students signed the Free Consent Term and Clarified (TCLE). The secrecy of the data collected in this study is kept absolutely reserved and used only for research purposes.

As for the risks of the intervention participants, they are minimal, as they are the same physical risks routinely encountered by students in physical education classes.

The activities will only be carried out by students who do not have physical or health limitations that could prevent physical activities. Any intercurrence of any risk to the student will be attended initially by the teacher in charge, in case of an emergency service, the Mobile Emergency Service System (SAMU) will be activated by contact phone 192. After the intervention, the student does not feel comfortable and wants to stop participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren from the 6th to the 9th grade of both sexes;
* Regularly enrolled in Full-time schools in the municipal public network of Canguçu/RS in the rural area;
* Have teachers with academic training in the field of Physical Education

Exclusion Criteria:

* Students who have disabilities or physical or cognitive limitations that prevent them from performing physical activities and/or compromise the answers to the questionnaires will be excluded from the study analysis. It is important to point out that if there is a student in this situation, they will participate normally in the intervention and measures (if they express their will and their guardians have consented), but their information will not be used.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cardiorespiratory Fitness | Cardiorespiratory Fitness will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  Cardiorespiratory fitness (m) will be measured based on performance in the six-minute run/walk test.
Change in Muscular Strength/Endurance | Muscular Strength/Endurance will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  Muscle strength/endurance (rep/min) will be evaluated by the number of sit-ups performed in one minute.
Change in Handgrip Strength | Handgrip Strength will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  The handgrip (kgf) strength will be evaluated by a handgrip dynamometer (Jamar®).
Change in Lower Limb Power | Lower limb power will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  Lower Limb Power (cm) will be evaluated by the horizontal jump test.
Change in Speed | Speed will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  Speed (s) will be assessed by the twenty meters sprint running test.
Change in Agility | Agility will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  Agility (s) will be assessed by the four by four meters square test.
Change in Flexibility | Flexibility will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  Flexibility (cm) will be assessed by the sit and reach test.
Change in Body Mass Index | Body Mass Index will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  Body Mass Index (kg/m2) will be calculated from the body mass (kg) and height (m) measures by the follow equation: body mass (kg) / height(m)2
Change in Waist Circunference | Waist Circunference will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  Waist Circunference (cm) will be measure using a flexible measuring tape with millimeter resolution positioned at the midpoint between the last rib and the iliac crest according to standardized procedures.
Change in Sum of Triceps and Subscapular Skinfolds | Sum of Triceps and Subscapular Skinfolds will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  Triceps and Subscapular Skinfolds (mm) will be measured by folding a double thickness of skin and adjacent adipose tissue, with index finger and thumb the fold must be pinched to facilitate the measurement and position the plicometer reader upwards according to standardized procedures.

SECONDARY OUTCOMES:
Changes in Physical Activity Level | Physical Activity Level will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  The level of physical activity (min/week) will be measured using the Physical Activity Questionnaire for Adolescents (QAFA).
Changes in Recreational Screen Time | Recreational Screen Time will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  Recreational screen time (min/day)will be assessed using the Questionnaire for Screen Time of Adolescents (QueST).
Changes in Sleep Time | Sleep Time will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  Sleep time (hours) will be measured through self-report considering the time that students indicate that they usually go to sleep and wake up on weekdays and weekends
Changes in Physical Self-Concept | Physical Self-Concept will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  Physical self-concept will be measured by the Physical Self-Concept Questionnaire wich is composed of 36 items divided into six factors: 1) PHYSICAL ABILITY; 2) PHYSICAL CONDITION; 3) PHYSICAL ATTRACTION; 4) STRENGTH; 5) GENERAL PHYSICAL SELF-CONCEPT; 6) GENERAL CONCEPT. For each factor, there are possible responses on a five-point Likert scale ("1-Strongly Disagree" - "5-Strongly Agree").
Changes in Motivation to Participate in Physical Education Classes | Motivation to Participate in Physical Education Classes will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  The motivation to participate in PE classes will be measured by the Perceived Locus of Causality Questionnaire (PLOCQ; Goudas et al., 1994) adapted and validated for the Brazilian reality by Tenório et al. (2019). The instrument consists of 20 questions based on the Theory of Self-Determination, being subdivided into five dimensions that assess different types of motivation, namely: intrinsic motivation, identified extrinsic motivation, introjected extrinsic motivation, external extrinsic motivation and amotivation, each consisting of for four items. For the response options, the Likert scale is used, with the following options: 1 - I strongly disagree; 2 - strongly disagree; 3 - disagree in general; 4 - neither agree nor disagree; 5 - I generally agree; 6 - strongly agree; 7 - I fully agree.
Changes in Symptoms of anxiety, depression and stress | Changes in Symptoms of anxiety, depression and stress will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  The symptoms of stress, anxiety and depression will be measured by the Depression Anxiety and Stress Scale (DASS-21) - Short Form, adapted and validated for Brazilian adolescents by Patias et al. (2016). This is a questionnaire reduced to 21 questions, seven for each item (stress, anxiety and depression). The evaluation of the aforementioned questionnaire is through a Likert-type scale with 4 scores: 0 It didn't happen to me this week; 1 It happened to me a few times a week; 2 It happened to me for most of the week; 3 It happened to me most of the time during the week. The sum of the answers (in each item and in the three items together) generates a score that can vary from zero (0) to twelve (12) for the items separately and thirty-six (36) for the three items together.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel G Bergmann, PhD, Principal Investigator — Escola Superior de Educação Física - Universidade Federal de Pelotas
Locations (1):
- Higher School of Physical Education - Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No